CLINICAL TRIAL: NCT01835795
Title: Prospective, Comparative, Randomized Study of the Effectiveness of Shock Wave Treatment in Myofascial Pain Syndrome in Low Back Pain
Brief Title: Radial Extracorporeal Shock Wave Treatment (rESWT) of Myofascial Pain Syndrome in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Kobayashi, Researcher and Collaborator of Pain Group, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 06251612.7.0000.0068
Record Dates: First submitted 2013-04-14; First posted 2013-04-19 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Myofascial Pain Syndromes; Low Back Pain; Lumbago
Keywords: Myofascial Pain Syndromes; Myofascial Trigger Point; Low Back Pain; Lumbago; Shock Waves, High-Energy; High-Energy Shock Waves; Interdisciplinary Health Team; Multidisciplinary Pain Centers
MeSH Terms: conditions — Myofascial Pain Syndromes; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radial Extracorporeal Shock Wave (Active Comparator): Swiss DolorClast® CLASSIC applicator
  Interventions: Device: Swiss DolorClast® CLASSIC applicator
- Placebo (Placebo Comparator): Swiss DolorClast® CLASSIC placebo applicator
  Interventions: Device: Swiss DolorClast® CLASSIC placebo applicator

INTERVENTIONS:
Device: Swiss DolorClast® CLASSIC applicator — Radial Extracorporeal Shock Wave applicator use in 6 sessions with 1 week of interval, 1000 impulses per myofascial trigger point, 5 to 7 hertz frequency, 2 to 4 bar pressure
  Arms: Radial Extracorporeal Shock Wave
Device: Swiss DolorClast® CLASSIC placebo applicator — Placebo applicator, use in 6 sessions with 1 week of interval, 1000 impulses per myofascial trigger point, 5 to 7 hertz frequency, 2 to 4 bar pressure
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of treatment of radial shockwave in myofascial pain syndrome in the lumbar region compared to placebo through questionnaires and imaging exams.

DETAILED DESCRIPTION:
BACKGROUND: Extracorporeal shockwave treatment has been used widely for musculoskeletal conditions, however no randomized controlled trial are available about its use for chronic low back pain with myofascial pain syndrome (MPS).

HYPOTHESIS: Radial extracorporeal shockwave treatment (rESWT) improves pain intensity and functional disability compared with placebo in patients with chronic low back pain due to MPS.

STUDY DESIGN: Randomized controlled clinical trial METHODS: A prospective, randomized, double-blind, placebo-controlled study will be carried out on 40 patients who has moderate to severe pain (VAS > 4) for more than 6 months, despite 6 weeks of conservative treatment with antidepressants associated with rehabilitation. Six interventions of rESWT (3-4 bar; 1000 impulses per trigger point (TP) or 2500 impulses per muscle) will be compared with placebo. The outcome measures were pain visual analogue scale (VAS), Oswestry Disability Index, Short-form McGill Pain Questionnaire, Roland Morris Disability Questionnaire and the temperature of the treated area will be evaluated with Thermography. The assessments will be apply before treatment, after conservative treatment, 6 and 12 weeks after rESWT.

ELIGIBILITY:
Inclusion Criteria:

* Presenting clinical complaints of lumbar and / or gluteal pains for 3 months or more
* Display pain of moderate to severe intensity: visual analogue scale (VAS)> 4
* Diagnosis of myofascial pain syndrome in the lumbar and / or gluteal
* Authorize in writing the term of free and informed consent to participate in the study
* Availability of frequent attendance at hospital

Exclusion Criteria:

* Organic or psychological disorders that contraindication participation of patients in study
* Metabolic, infectious, oncological or rheumatologic disorders
* Fibromyalgia
* Labor dispute
* Indication for surgery in column
* Contraindications to therapy of shock waves:

  * Coagulopathy and / or anticoagulant
  * Pregnancy
  * Acute infection in soft tissue or bone
  * Systemic Infections
  * Presence of ulcers at treatment sites
  * Presence of larger vessels or nerves at treatment sites
  * Polyneuropathies
  * Malignancies
  * Cardiac arrhythmias or use of pacemaker
  * Epilepsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Evidence of pain relief by visual analogue scale (VAS) of radial extracorporeal shock waves in myofascial pain syndrome in the lumbar and gluteal region compared to placebo | 12 weeks after the last session of shockwave
  The outcome will be assessed by Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Kobayashi, Principal Investigator — IOT HCFMUSP - Instituto de Ortopedia e Traumatologia do Hospital das Clínicas da Faculdade de Medicina da USP
Locations (1):
- IOT HCFMUSP - Instituto de Ortopedia e Traumatologia do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil